CLINICAL TRIAL: NCT05550740
Title: Repeated Low-Level Red-Light Therapy for Shortening Axial Length in Chinese High Myopia Children and Teenagers: a Prospective Single-Arm Study
Brief Title: Repeated Low-Level Red-Light Therapy for Shortening Axial Length
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMRL-SEPTC-2022
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-11

CONDITIONS: High Myopia; Refractive Errors; Eye Diseases
MeSH Terms: conditions — Refractive Errors; Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RLRL therapy (Experimental): In addition to SVS, participants will be treated with RLRL twice a school day.
  Interventions: Device: RLRL

INTERVENTIONS:
Device: RLRL — In addition to SVS with power for correcting distance refraction, RLRL will be performed twice per school day with an interval of at least 4 hours, each treatment last 3 minutes.

SUMMARY:
The purpose of this clinical trial is to confirm the incidence and magnitude of axial length shortening after RLRL therapy in Chinese high myopia children and teenagers.

DETAILED DESCRIPTION:
High myopia has become a major public concern globally, which is characterized by excessive axial elongation of the eyeball. Axial elongation is accompanied by mechanical stretching and thinning of the choroid and sclera, causing vision-threatening complications. RLRL therapy is an emerging effective and safe therapy for myopia control. Previous clinical trials in China have observed clinically significant axial shortening after RLRL treatment.

The purpose of this study is to confirm and identify possible mechanism for axial length (AL) shortening after 12-month RLRL therapy in Chinese highly myopic children and teenagers aged 6-16 years. In addition to single vision spectacles, subjects will receive RLRL treatment at home under supervision of the parents according to a standard protocol. Axial length, visual acuity, cycloplegic spherical equivalent refraction, intraocular pressure, slit lamp, optical coherence tomography, optical coherence tomography angiography and ultrawide-field optical coherence tomography will be measured at 1-, 3-, 6- and 12-month follow-up visits. This trial will be extended to 3 years and follow-up visits are scheduled at 18-, 24-, 30- and 36-month.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of consent.
2. Age: ≥ 6 and ≤ 16 years at enrolment.
3. High myopia: cycloplegic sphere ≤ -6.00 diopters (D) in both eyes.
4. Willing and able to participate in all required activities of the study.
5. The children currently on myopia control treatment can be recruited if myopia control treatments (including but not limited to atropine, orthokeratology, rigid gas-permeable lenses, defocus spectacles, etc.) are discontinued for at least 2 weeks.
6. Normal fundus, tessellated fundus or with peripapillary diffuse chorioretinal atrophy.

Exclusion Criteria:

1. Secondary myopia, such as a history of retinopathy of prematurity or neonatal problems, or syndromic myopia with a known genetic disease or connective tissue disorders, such as Stickler or Marfan syndrome.
2. Pathologic myopia with signs of macula-involving diffuse chorioretinal atrophy, patchy chorioretinal atrophy, macular atrophy, lacquer cracks, myopic choroidal neovascularization or Fuchs' spots.
3. Strabismus and binocular vision abnormalities in either eye.
4. Previous any intraocular surgery affecting refractive status.
5. Other reasons, including but not limited to ocular or other systemic abnormalities, that the physician may consider inappropriate for enrolment.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-11-19 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Incidence rate (%) of axial length shortening >0.05 mm measured by the IOL Master | 12 months
  Incidence rate of axial length shortening > 0.05 mm is characterized as the ratio of number of participants with axial length shortening greater than 0.05 mm to the total number.

SECONDARY OUTCOMES:
Incidence rates (%) of axial length shortening >0.10 mm and >0.20 mm measured by the IOL Master | 12 months
  Incidence rate of axial length shortening > 0.10 mm and 0.20 mm are characterized as the ratio of number of participants with axial length hortening greater than 0.10 mm and 0.20 mm to the total number.
Changes of axial length shortening (mm) among shortened eyes measured the IOL master | 12 months
  Changes of axial length shortening is characterized as the magnitude of axial length reduction among axial shortened eyes.
Changes in choroidal structural and perfusion parameters measured by the swept-source optical coherence tomography and optical coherence tomography angiography | 1, 3, 6 and 12 months
  Changes in choroidal structural and perfusion parameters are characterized as the difference between each follow-up visit and corresponding baseline values. Indicators include choroidal vascular index, choroidal thickness and so on.
Changes in retinal structures by the swept-source optical coherence tomography and optical coherence tomography angiography | 1, 3, 6 and 12 months
  Swept-source optical coherence tomography is used to measure retinal structures. The structures of nerve sensory layer, retinal pigment epithelium layer and choroid layer were observed by fundus images.
Changes in axial length (mm) and other biometric parameters (mm, μm) by the IOL master | 1, 3, 6 and 12 months
  The IOL Master is used to measure axial length and other biometric parameters, including corneal curvature, anterior chamber depth and white to white, etc. Change of each parameter is characterized as the difference between each follow-up visit and baseline values
Change of cycloplegic spherical equivalent refraction (Diopter) by the autorefractor | 1, 3, 6 and 12 months
  Cycloplegic spherical equivalent change (Diopter, D) is characterized as the difference between each follow-up visit and baseline values. Refraction with full cycloplegia is performed with an autorefractor. The data on spherical and cylindrical power and axis is automatically extracted from the autorefractor. The spherical equivalent power (D) is calculated as the spherical power (D) plus half of the cylindrical power (D)
Change of pathologic myopia fundus META-PM grading | 1, 3, 6 and 12 months
  The swept-source optical coherence tomography is used to obtain fundus images. The fundus images are classified based on META-PM classification system
Change in best corrected visual acuity (logMAR) by the Early Treatment Diabetic Retinopathy Study (ETDRS) logMAR chart | 1, 3, 6, and 12 months
  Best corrected visual acuity change is characterized as the difference between each follow-up visit and baseline values. An Early Treatment Diabetic Retinopathy Study chart with standard illumination at a distance of 4 meters is used to measure best corrected visual acuity
Incidence (%) of self-reported adverse events by the quesionnaire including but not limited to glare, flash blindness, and afterimages | 1, 3, 6 and 12 months
  Incidence of self-reported adverse events is the rate of self-reported adverse events over a specified period for all the subjects.

OTHER OUTCOMES:
Full myopia control rate (%) by the autorefractor | 36 months
  Cycloplegic spherical equivalent change (Diopter, D) is characterized as the difference between each follow-up visit and baseline values. Refraction with full cycloplegia is performed with an autorefractor. The data on spherical and cylindrical power and axis is automatically extracted from the autorefractor. The spherical equivalent power (D) is calculated as the spherical power (D) plus half of the cylindrical power (D). Full myopia control is defined as cycloplegic SER progression <0.25 D/year.
Morphological changes of the posterior ocular segment by the quantitative ultrawide-field optical coherence tomography | 36 months
  Morphological changes of the posterior ocular segment is measured using the quantitative ultrawide-field optical coherence tomography between follow-up visit and baseline.
Changes in axial length (mm) and other biometric parameters (mm, μm) by the IOL master | 36 months
  The IOL Master is used to measure axial length and other biometric parameters, including corneal curvature, anterior chamber depth and white to white. Change of each parameter is characterized as the difference between each follow-up visit and baseline values.
Changes in choroidal structural and perfusion parameters measured by the swept-source optical coherence tomography and optical coherence tomography angiography | 36 months
  Changes in choroidal structural and perfusion parameters are characterized as the difference between each follow-up visit and corresponding baseline values. Indicators include choroidal vascular index, choroidal thickness and so on.
Change in visual acuity (logMAR) by the Early Treatment Diabetic Retinopathy Study (ETDRS) logMAR chart | 36 months
  Visual acuity change is characterized as the difference between each follow-up visit and baseline values. An ETDRS chart with standard illumination at a distance of 4 meters is used to measure visual acuity.
Incidence (%) of self-reported adverse events by the quesionnaire including but not limited to glare, flash blindness, and afterimages | 36 months
  Incidence of self-reported adverse events is the rate of self-reported adverse events over a specified period for all the subjects. Subjects are asked to report any treatment-emergent adverse events, including but not limited to glare, flash blindness, and afterimages.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention and Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared as open data after proper anonymization.